CLINICAL TRIAL: NCT04894500
Title: The Intensive Care Infection Score in Adult and Paediatric Burns in Comparison to Other Inflammatory Markers
Brief Title: ICIS in Burn Patients Compared to Other Inflammatory Markers
Acronym: ICARUS
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Bohumil Bakalar MD, Intensive Care lead, Charles University, Czech Republic
Other Study IDs: 0402021
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2023-08

CONDITIONS: Infection, Bacterial; Burns; Inflammation
MeSH Terms: conditions — Bacterial Infections; Burns; Inflammation | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flow fluorescence cytometry — Level of inflammatory markers in body fluid samples
  Other Names: CRP; PCT; Presepsin; IL-6; TNF-α; WBC

SUMMARY:
The current markers of inflammation that govern antibiotic treatment have their significant limitations, especially in patients with burns. According to previously published data, the newly proposed marker of infectious inflammation, the Intensive Care Infection Score (ICIS), appears to be a suitable diagnostic tool in distinguishing between inflammation of infectious and non-infectious origin in these patients. The other advantage is its low price.

This study aims to compare ICIS with other used indicators of inflammation in patients with burns both children and adults.

DETAILED DESCRIPTION:
Improving the use of antibiotics is an important patient and public health issue. The misuse of antibiotics has contributed to the growing problem of antibiotic resistance, which has become one of the most serious and growing threats to public health.

The prompt initiation of antibiotics to treat infections has been proven to reduce morbidity and save lives, however, up to 30% of all antibiotics prescribed in ITUs are either unnecessary or inappropriate. One of the key problems is early and reliable detection of infection. Specificity of clinical signs and routine laboratory markers is low and they usually cannot distinguish among changes caused by the primary insult, inflammatory reaction, and infection.

The gold standard of systemic bacterial and fungal infection, i.e. positive blood culture, has a sensitivity of less than 75 per cent and its contamination has been found in up to one third of results. Sputum and urine cultures are contaminated even more. Moreover, culture results are usually not known earlier than after 48 hours and antibiotic treatment should be started earlier in many cases, especially in the case of septic shock.

New diagnostic modalities have been developed to sort out difficulties with early and reliable diagnosis of a presence of infection, for example measurement of Procalcitonin (PCT) or Presepsin level, matrix-assisted laser desorption ionization time-of-flight detector mass spectrometry (MALDI TOF MS), DNA hybridisation, and polymerase chain reaction (PCR) tests, eventually polymerase chain reaction electrospray ionization mass spectrometry (PCR ESI-MS).

PCT examination is the most used laboratory test from the modalities mentioned above. Despite many positive characteristics (i.e. fast dynamics of plasma changes, higher sensitivity and specificity than C-reactive protein, ability to distinguish between G+ and G- infection), PCT specificity drops in patients with ARDS, burns, multiple injuries, rhabdomyolysis, lysis of lymphocytes, extreme metabolic situations, organ perfusion failure and after large surgical procedures. It is also worth mentioning the relatively high cost of this examination, limiting the use of this marker for routine screening, especially in low- and middle-income countries.

The limiting factor for the use of the other diagnostic methods mentioned above is their availability and price, or the fact that they are not reimbursed by health insurance companies. Thus, the need for a reliable, cost-effective and available marker to facilitate antibiotic therapy continues to be a burning problem, especially in intensive care, where the development of SIRS is part of the disease in many patients.

Intensive Care Infection Score (ICIS) has been proposed as a suitable diagnostic indicator for the presence of infection in these patients. Five parameters are used to calculate this score:

* Number of neutrophil segments
* The number of immature granulocytes
* Mean fluorescence intensity of neutrophil segments
* Difference in haemoglobin concentration of mature and young cells
* Number of antibody secreting lymphocytes These parameters characterize the early innate immune response. The maximum ICIS value is 20. ICIS changes occur in the order of hours and are capable of detecting early local and systemic infection prior to the development of clinical symptoms. The advantages are the low cost of the examination which can be used to routinely screen patients, the speed of results (up to 15 min), sensitivity, assessment of the severity of infection, and the fact that no extra blood sample is needed. Measurements are done from a blood sample taken for differential blood count by flow fluorescence cytometry.

Nevertheless, ICIS suitability and accurance in both adult and pediatric burn patients has not been proved yet. This study is aimed to investigate ICIS reliability in burns.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized on Prague Burn Centre, Czech Republic, for more than 3 days.

Exclusion Criteria:

* Refusal to sign informed consent or withdrawal of already signed consent;
* Patient in palliative care.

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted for burn injuries.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The Intensive Care Infection Score is not inferior to selected inflammatory markers in detection of bacterial infection | 15 days
  Comparison of the ICIS to CRP, PCT, IL-6, WBC, TNF-α, and Presepsin

SECONDARY OUTCOMES:
The Intensive Care Infection Score is a suitable biomarker for distinguishing bacterial infection from systemic inflammatory response syndrome (SIRS) | 30 days
  Comparison of the ICIS to microbial results
The Intensive Care Infection Score does not depend on the extend and depth of the burn area | 5 days
  Comparison of the ICIS and burn characteristics
The Intensive Care Infection Score is a suitable marker of bacterial infection in children with burns | 10 days
  Suitability of the ICIS in pediatric patients with thermic injury

CONTACTS AND LOCATIONS:
Overall Officials: Helena Lahoda Brodská, MD, PhD, Principal Investigator — Ústav lékařské biochemie a laboratorní diagnostiky 1. LF UK a Všeobecné fakultní nemocnice Praha
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
We plan to allow access to a database created on Google

REFERENCES:
- [Background] van der Geest PJ, Mohseni M, Linssen J, Duran S, de Jonge R, Groeneveld AB. The intensive care infection score - a novel marker for the prediction of infection and its severity. Crit Care. 2016 Jul 7;20(1):180. doi: 10.1186/s13054-016-1366-6. PMID 27384242
- [Background] Nierhaus A, Linssen J, Wichmann D, Braune S, Kluge S. Use of a weighted, automated analysis of the differential blood count to differentiate sepsis from non-infectious systemic inflammation: the intensive care infection score (ICIS). Inflamm Allergy Drug Targets. 2012 Apr;11(2):109-15. doi: 10.2174/187152812800392841. PMID 22280231
- [Background] Weimann K, Zimmermann M, Spies CD, Wernecke KD, Vicherek O, Nachtigall I, Tafelski S, Weimann A. Intensive Care Infection Score--A new approach to distinguish between infectious and noninfectious processes in intensive care and medicosurgical patients. J Int Med Res. 2015 Jun;43(3):435-51. doi: 10.1177/0300060514557711. Epub 2015 Apr 7. PMID 25850686